CLINICAL TRIAL: NCT04724824
Title: Validation of a Brain-Computer Interface for Neurorehabilitation With a Randomized Controlled Trial (Validación de Una Interfaz Cerebro-Computadora Para Rehabilitación Neurológica Por Medio de un Ensayo Clínico Controlado y Aleatorizado)
Brief Title: Validation of a Brain-Computer Interface for Stroke Neurological Upper Limb Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other); Hospital General Dr. Manuel Gea González (Other Government); El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Responsible Party: Principal Investigator, Jessica Cantillo-Negrete, Researcher in Medical Sciences, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SALUD-2018-02-B-S-45803
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Stroke, Ischemic; Stroke
Keywords: brain-computer interface; robotic orthosis; hemiparesis; motor rehabilitation
MeSH Terms: conditions — Ischemic Stroke; Stroke; Paresis | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain-Computer Interface controlled robotic feedback (Experimental)
  Interventions: Device: Brain-Computer Interface
- Sham Brain-Computer Interface controlled robotic feedback (Sham Comparator)
  Interventions: Device: Sham Brain-Computer Interface

INTERVENTIONS:
Device: Brain-Computer Interface — Passive hand movement will be provided to patients' paralyzed hand by means of a robotic hand orthosis that will be activated by the brain-computer interface based on hand movement intention.
  Arms: Brain-Computer Interface controlled robotic feedback
Device: Sham Brain-Computer Interface — Passive hand movement will be provided to patients' paralyzed hand by means of a robotic hand orthosis which activation will be independent of the output of the brain-computer interface based on hand movement intention.
  Arms: Sham Brain-Computer Interface controlled robotic feedback

SUMMARY:
The study's main goal is to determine if clinical and physiological effects of a brain-computer interface intervention for the neurorehabilitation of stroke patients' upper limb are greater than the effects of a sham robotic feedback. For this purpose a randomized controlled trial will be performed to compare somatosensory sham robotic feedback with the same somatosensory feedback controlled with the brain-computer interface output.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of first ischemic stroke
* Time since stroke onset higher than 3 months and lower than 24 months
* Hand paresis
* Normal or corrected to normal vision
* Without previous diagnosed neurological diseases

Exclusion Criteria:

* Clinical diagnosis of severe aphasia
* Clinical diagnosis of severe depression
* Clinical diagnosis of severe attention deficits
* Previous diagnosis of traumatic brain injury
* Previous diagnosis of spinal cord injury
* Previous diagnosis of peripheral nerve injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in upper limb motor function on the Fugl-Meyer Assessment for the Upper Extremity | At enrollment, 3 weeks after the intervention onset, 6 weeks after the intervention onset, and 24 weeks after the intervention onset
  Analysis of changes on the Fugl-Meyer Assessment for the Upper Extremity will reveal if there is a clinical significant sensorimotor function compared to baseline
Mean change from baseline in upper limb motor function on the Action Research Arm Test | At enrollment, 3 weeks after the intervention onset, 6 weeks after the intervention onset, and 24 weeks after the intervention onset
  Analysis of changes on the Action Research Arm Test will reveal if there is a clinical significant motor function compared to baseline

SECONDARY OUTCOMES:
Mean change from baseline in cortical activity measured with Functional Magnetic Resonance Imaging | At enrollment, 3 weeks after the intervention onset, 6 weeks after the intervention onset, and 24 weeks after the intervention onset
  Blood-oxygen-level-dependent imaging will be analyzed to assess if there are changes in cortical activity compared to baseline.
Mean change from baseline in corticospinal excitability measured with Transcranial Magnetic Stimulation | At enrollment, 3 weeks after the intervention onset, 6 weeks after the intervention onset, and 24 weeks after the intervention onset
  Motor Evoked Potentials parameters will reveal if there are changes of corticospinal excitability in both hemibodies compared to baseline
Mean change from baseline in grip strength measured with a dynamometer | At enrollment, 3 weeks after the intervention onset, 6 weeks after the intervention onset, and 24 weeks after the intervention onset
  Analysis of hand strength measurements will reveal if there were changes compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Cantillo-Negrete, PhD, Principal Investigator — Instituto Nacional de Rehabilitacion (National Institute of Rehabilitation)
Locations (1):
- Instituto Nacional de Rehabilitacion Luis Guillermo Ibarra Ibarra (National Institute of Rehabilitation), Tlalpan, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected during the study will be available to other researchers from the principal investigator on reasonable request.
Supporting Information: CSR
Time Frame: Six months after publication
Access Criteria: Researchers that make a request for access data and their request is approved by the National Institute of Rehabilitation Ethics Committee

REFERENCES:
- [Derived] Cantillo-Negrete J, Rodriguez-Garcia ME, Carrillo-Mora P, Arias-Carrion O, Ortega-Robles E, Galicia-Alvarado MA, Valdes-Cristerna R, Ramirez-Nava AG, Hernandez-Arenas C, Quinzanos-Fresnedo J, Pacheco-Gallegos MDR, Marin-Arriaga N, Carino-Escobar RI. The ReHand-BCI trial: a randomized controlled trial of a brain-computer interface for upper extremity stroke neurorehabilitation. Front Neurosci. 2025 Jun 18;19:1579988. doi: 10.3389/fnins.2025.1579988. eCollection 2025. PMID 40606836
- [Derived] Rodriguez-Garcia ME, Carino-Escobar RI, Carrillo-Mora P, Hernandez-Arenas C, Ramirez-Nava AG, Pacheco-Gallegos MDR, Valdes-Cristerna R, Cantillo-Negrete J. Neuroplasticity changes in cortical activity, grey matter, and white matter of stroke patients after upper extremity motor rehabilitation via a brain-computer interface therapy program. J Neural Eng. 2025 Mar 20;22(2). doi: 10.1088/1741-2552/adbebf. PMID 40064104